CLINICAL TRIAL: NCT02776202
Title: HLA-Identical Sibling Donor Bone Marrow Transplantation for Individuals With Severe Sickle Cell Disease Using a Reduced Intensity Conditioning Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC15/043/R
Record Dates: First submitted 2016-05-15; First posted 2016-05-18 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — fludarabine phosphate; Melphalan; Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced-intensity conditioning regimen (Experimental): The HSCT preparative regimen will consist of
  * Thymoglobulin: 2.5 mg /kg/day intravenously (IV) on Days -8 through -5
  * Fludarabine: 35 mg/m2/day IV on Days -8 through -4
  * Melphalan: 140 mg/m2 IV on Day -3
  * Rest on Day -2 and -1
  * Day 0 is the day of transplant
  * GVHD prophylaxis: sirolimus beginning on Day -1 for at least one year and mycophenolate mofetil (MMF) from Day -3 to +45 or to 7 days after neutrophil engraftment, whichever is later.
  Interventions: Drug: Fludarabine monophosphate

INTERVENTIONS:
Drug: Fludarabine monophosphate — The HSCT preparative regimen will consist of
  * Thymoglobulin: 2.5 mg /kg/day intravenously (IV) on Days -8 through -5
  * Fludarabine: 35 mg/m2/day IV on Days -8 through -4
  * Melphalan: 140 mg/m2 IV on Day -3
  * Rest on Day -2 and -1
  * Day 0 is the day of transplant
  * GVHD prophylaxis: sirolimus beginning on Day -1 for at least one year and mycophenolate mofetil (MMF) from Day -3 to +45 or to 7 days after neutrophil engraftment, whichever is later.
  Other Names: Melphalan; Mycophenolate Mofetil; Sirolimus

SUMMARY:
Sickle cell disease (SCD) is the most common inherited blood disorder in Saudi Arabia . Its clinical severity is widely heterogeneous among patients who share the same genetic mutation . Severe frequent pain crisis, recurrent acute chest syndrome and stroke are features of severe SCD. Hydroxyurea is an effective treatment of SCD as it ameliorates the severity and frequency of pain crisis and acute chest syndrome and decreases mortality, however, it is less effective in the prevention and treatment of stroke and other end organ dysfunctions . The only readily available cure of SCD is by hematopoietic stem cell transplantation (HSCT) . Most children with SCD who are treated by HSCT receive myeloablative conditioning with excellent results. The application of reduced intensity (RIC) and non-myeloablative (NMA) conditioning regimens are reserved for patients older than 16 years of age because of the increased risks of morbidity and mortality after HSCT6. However, infertility and gonadal failure after myeloablative conditioning are important barriers to the willingness of patients and their families to undergo HSCT . The development of an effective RIC HSCT in SCD that might spare the fertility of SCD patients would have obvious merit.

With the ultimate goal of expanding this curative therapy to SCD patients, we propose to investigate HSCT with a RIC conditioning regimen. We will carry out a pilot study of HSCT from HLA matched sibling donors using thymoglobulin/fludarabine/melphalan conditioning and sirolimus and mycophenolate mofetil (MMF) as GVHD prophylaxis in SCD patients with severe complications such as stroke and other severe complications. We hypothesize that HSCT from HLA matched sibling using thymoglobulin/fludarabine/melphalan conditioning in SCD will maintain a level of stable donor chimerism that is sufficient to cure SCD with minimal toxicity.

DETAILED DESCRIPTION:
Busulfan-based myeloablative allogeneic HSCT from an HLA-matched related donor in children is associated with high cure rate ranging from 80-90% in different trials, reviewed in 6. Lessons learned from these trials include; rabbit ATG significantly contributes to a lower graft rejection rate, the presence of stable mixed chimerism is sufficient to cure SCD, and the risk of neurological toxicities was minimized by maintaining platelet count greater than 50,000/uL and hemoglobin level between 9-11g/dL, adding phenytoin prophylaxis, and preventing hypertension and hypomagnesemia . We will not present results of these trials here, as the focus of this proposal is to investigate the use of NMA/RIC HSCT in SCD.

2.1 RIC/NMA HSCT in SCD:

1. Van Besien et al 8 reported transplant results in two adults with SCD who underwent allogeneic transplantation from an HLA-identical sibling donor after conditioning with fludarabine/melphalan and ATG. One patient was a 40-year-old female who had significant end-organ dysfunction related to SCD (renal failure treated by dialysis, pulmonary diffusion capacity was reduced by 25% and ischemic stroke) and was heavily transfused prior to transplant. She also had RBC alloantibodies and was receiving hydroxyurea and erythropoietin. She was conditioned with ATG 30 mg/kg for 4 consecutive days (day -5 to day -2), fludarabine 30 mg/m2 i.v. for 4 consecutive days (day -5 to day -2) and melphalan 140 mg/m2 i.v. on day -1. The patient had hemodialysis performed on day -5, day -3 and day -1 after chemotherapy was administered. On day 0, the patient received an infusion of cryopreserved G-CSF-mobilized peripheral blood stem cells (PBSC). GVHD prophylaxis consisted of daily tacrolimus and mini methotrexate regimen (5 mg/m2 given on days 1, 3 and 6). There was successful neutrophil and platelet engraftment and 100% stable chimerism. She developed interstitial pneumonia, possibly secondary to GVHD, 140 days after transplantation and progressed to respiratory failure leading to her death on day 355. The second patient was a 56 year old with SC disease who was heavily pretransfused and had multiple SCD complications. She received the same conditioning, GVHD prophylaxis, and PBSC source as the first patient. She had 100% donor chimerism but died on day 142 secondary to TTP and severe gut GVHD with CNS infection.
2. Iannone et al 9 described 6 pediatric patients with SCD who underwent bone marrow transplant from their HLA matched siblings after conditioning with fludarabine 50mg/m2/day for 3-5 days and 200 cGy TBI in addition to horse ATG in one patient. GVHD prophylaxis included MMF and tacrolimus or cyclosporine with various taper schedules. There was minimal toxicity, however, all patients developed graft rejection upon taper of immunosuppressive medications.
3. Horan et al 10 described three SCD patients who were heavily transfused prior to transplant and underwent HLA matched sibling transplant after conditioning with fludarabine 25mg/m2 on 5 consecutive days before transplantation (days -6 to -2), rabbit ATG (Thymoglobulin) on 4 consecutive days before transplantation (days -6 to -2) with age adjusted dose, and single dose TBI 200 cGy. GVHD prophylaxis included MMF in the first three months and CSA for at least six months. All had graft rejection except one when the immunosuppression was tapered. There was no GVHD.
4. Horwitz et al 11 reported the outcome in two adult SCD patients who underwent HLA matched sibling transplant and PBSC was the source of graft in both cases. Conditioning was TBI 200 cGy followed by fludrabine 24-30 mg/m2 for 4 days and cyclophosphamide 500 mg/m2 for four days and alemtuzumab 100mg for five days. MMF was given in the first 100 days post transplant. Both engrafted successfully with no GVHD and a follow up of 20 months.
5. Krishnamurti et al described the use of RIC in seven SCD patients, age range 6-16 years. The conditioning was busulfan 3.2 mg/kg on day -8 and -7, fludarabine 35mg/m2 on days -6 to -2, equine ATG 30mg/kg on days -5 to -1, and total lymphoid irradiation. GVHD prophylaxis was CSA and MMF. CSA was tapered starting day +180 and MMF taper varied from +45 to +220 day. Six patients had stable mixed chimerism after stopping CSA and MMF. One patient had late graft failure. There was a low rate of GVHD.
6. Hsieh et al reported the use of non-myeloablative conditioning in SCD patients older than 16 years of age. Graft source was GCSF mobilized PBSC from HLA matched siblings with at least 10 X106 CD34/kg of recipient weight. Conditioning was alemtuzumab (total 1mg/kg divided on days -7 to -3) and single dose TBI 300 cGy on day -2. Presence of major ABO incompatibility was one of the exclusion criteria for this study. Sirolimus was used as GVHD prophylaxis and to prevent graft rejection. Nine of 10 patients engrafted successfully and had stable chimerism, however, all patients continue to be on sirolimus. None of patients had GVHD. They recently updated these promising results in a total of 30 patients and were able to taper off sirolimus in 15 patients.

2.2 Rationale for using thymoglobulin/fludarabine/melphalan conditioning RIC is a feasible option for patients with SCD and can successfully cure the disease. A pre-transplant backbone regimen consisting of Alemtuzumab or ATG, fludarabine, and melphalan has been applied successfully in SCD patients as described above. We anticipate that the toxicity risk is lower than the full myeloablative conditioning using busulfan and cyclophosphamide (BU/CY). Melphalan was reported to cause infertility, mostly when we used with other chemotherapy agents. The use of melphalan alone in the conditioning regimen was reported before to potentially preserve fertility in women. So our regimen could potentially preserve fertility at higher rate compared to BU/CY.

2.3 Rationale for pre-transplant immunosuppression therapy with hydroxyurea Individuals with hemoglobinopathies have in general adequate T cell function and active bone marrow that can lead to higher risk of graft rejection especially among patients who are heavily transfused. Experience with class 3 thalassemia patients showed that pretreatment with hydroxyurea, azathioprine, and fludarabine decreased the risk of graft rejection and allowed the use of lower dose cyclophosphamide . So we will use hydroxyurea prior to transplant to minimize the risk of graft rejection associated with RIC in sickle cell anemia.

2.4 Rationale for using sirolimus and MMF as GVHD prophylaxis: Post-grafting immunosuppression appears crucial to ensuring stable engraftment; an early taper appears to contribute to late graft rejection in several of the series. Sirolimus is an inhibitor of the mammalian target of rapamycin (mTOR) and it induces immune tolerance and was used successfully as GVHD prophylaxis in adult SCA patients who underwent RIC/ NMA. Sirolimus in combination with calcineurin inhibitors or MMF was utilized effectively in pediatric patients 19-21. However, studies showed increased risk of veno-occlusive disease with the combination of sirolimus and MMF and increased risk of transplant-associated thrombotic microangiopathy when combined with tacrolimus especially among patients who received busulfan-based conditioning 22-24. We will be using a RIC regimen so we do not anticipate that the combination of sirolimus and MMF will cause excess toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 1. SCD patients who are 3-18 years old. 2. SCD (HbSS, HbSβ° thalassemia or any genotype) with at least one of the following conditions:

  1. Clinically significant neurologic event (stroke) or any neurologic defect lasting > 24 hours and accompanied by an infarct on cerebral magnetic resonance imaging (MRI)
  2. Minimum of two episodes of acute chest syndrome within the preceding 2-year period defined as new pulmonary alveolar consolidation involving at least one complete lung segment (associated with acute symptoms including fever, chest pain, tachypnea, wheezing, rales or cough that is not attributed to asthma or bronchiolitis) despite adequate supportive care measures
  3. History of 3 or more severe pain events per year in the 2 years prior to enrollment.

     3. Availability of 10/10 genotypically HLA identical related donor 4. In patients who have been treated by regular RBC transfusions >12 months, with a liver biopsy that shows no evidence of cirrhosis or active hepatitis 5. Patients must have a Karnofsky score ≥ 50 or WHO/ECOG ≥ 2 for patients age ≥ 16, Lansky score ≥ 50 for patients age < 16.

     6. Adequate cardiac function: shortening fraction of > 25% or ejection fraction of > 55% by echocardiogram 7. Adequate renal function: serum creatinine within normal limits or creatinine clearance >70 ml/min/1.73 m2 8. Adequate liver function: Total bilirubin within normal limits and AST/ALT <2.5x upper limit of normal

     Exclusion Criteria:
* 1. Patients with symptomatic cardiac insufficiency or arrhythmia. 2. Patients with cirrhosis on liver biopsy. 3. Hepatitis B, hepatitis C, or HIV seropositive patients. 4. Patients with other disease that would increase toxicity of transplant.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
to determine event-free survival (EFS) at 1 year after HLA-Identical sibling donor hematopoietic stem cell transplantation (HCT) using bone marrow (BM) in patients with sickle cell disease (SCD). | 3 years

SECONDARY OUTCOMES:
1. To determine the effect of HCT on clinical and laboratory manifestations of severe sickle cell disease including stroke. | 3 years
determine the incidence of other transplant-related outcomes. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdul Aziz Medical City for National Guard, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided